CLINICAL TRIAL: NCT06509542
Title: Measuring the Concurrent Validity of the Upper Limb Use Ratio With Accelerometers in an Ecological Situation After Stroke. ValidFUR
Brief Title: Measuring the Concurrent Validity of the Upper Limb Use Ratio With Accelerometers in an Ecological Situation After Stroke.
Acronym: ValidFUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Paul Coste Floret Hospital (Unknown); Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0428
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Cerebrovascular Accident
Keywords: Learned non-use; Accelerometer; Neurorehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: While patients are in rehabilitation, upper limb movements will be recorded using wrist-worn accelerometers and video cameras, during dressing, meal preparation, and meal-taking activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measure of FuncUseRatio using wrist-worn accelerometers and videos (Experimental): The wristbands are made from hypoallergenic silicone and weigh 27 grams. They contain three accelerometers (AX3, Axivity, Newcastle Helix, United Kingdom), recording data in the three planes of space at a sampling frequency of 50 Hz and within an acceleration range of ±8 g. The wristbands will be worn on each wrist during the activities.
  Two high-definition video cameras, recording at least 50 images per second, will be positioned so that the movements of the patient's upper limbs are always visible. The location of the cameras will depend on the activity and the configuration of the room in which it takes place.
  Interventions: Behavioral: Objective assessment of upper limb use during activities in ecological situation

INTERVENTIONS:
Behavioral: Objective assessment of upper limb use during activities in ecological situation — Twenty-five patients will be recorded performing three activities during their rehabilitation: getting dressed, preparing a meal, and eating a meal. The movements of their upper limbs will be tracked using wrist-worn accelerometers and video cameras.

SUMMARY:
The purpose of this stufy is to measure the concurrent validity of the upper limb use ratio with accelerometers in an ecological situation after stroke.

DETAILED DESCRIPTION:
The first visit will be used to present the study and potential risks to patients, obtain their consent and collect clinical data. A second visit is planned for the patients who meet the eligibility requirements, to carry out activities in ecological situation.

ELIGIBILITY:
Inclusion Criteria:

* Subject with hemiparesis following stroke
* Subject participating in ecological activities during occupational therapy sessions
* Adult subject aged 18 or over
* Subject informed of study participation and not objecting to participation

Exclusion Criteria:

* Other neurological or musculoskeletal disorders limiting use of upper limbs
* Pregnant or breast-feeding woman,
* Failure to obtain consent,
* Non-affiliation with a social security scheme,
* Persons under court protection,
* Person protected by law (under guardianship or curatorship)
* Participant in another research project with an exclusion period still ongoing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Concurrent validity (Intraclass Correlation Coefficient) of FuncUseRatio, using wrist-worn accelerometers, compared with the FuncUseRatio measured by video analysis. | Baseline
  FuncUseRatio is the ratio of functional use of the paretic upper arm to the non-paretic upper arm measured by two methods (actimetry and video analysis),during the same occupational therapy sessions simulating activities of daily living with hemiparetic patients.

SECONDARY OUTCOMES:
Number of functional movements performed with the upper limbs (FuncUse30) | Baseline
  The functional movements are the movements with an amplitude greater than 30° within a spatial range of -30° to +30° around the horizontal, measured over a two-second time window (FuncUse30)
Ratio of the acceleration vector magnitude | Baseline
  The magnitude of the acceleration vector is the norm of the acceleration vector (SVM: Scalar Vector Magnitude) minus 1 for the gravitational force. The ratio between the paretic and non paretic arm is then calculated
Activity count ratio | Baseline
  The activity count is the magnitude of the acceleration vector summed per second for each arm, and converted into an activity count (0.01664g/count). The ratio between the paretic and the non-paretic arm is then calculated.
Activity time ratio | Baseline
  The activity time is the sum of the seconds of arm activity for each arm. The ratio between the paretic and the non-paretic arm is then calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH Paul Coste Floret, Lamalou-les-Bains
  - CHU Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faity G, Mottet D, Pla S, Froger J. The reserve of joint torque determines movement coordination. Sci Rep. 2021 Nov 26;11(1):23008. doi: 10.1038/s41598-021-02338-4. PMID 34836976
- [Result] Bailey RR, Klaesner JW, Lang CE. Quantifying Real-World Upper-Limb Activity in Nondisabled Adults and Adults With Chronic Stroke. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):969-78. doi: 10.1177/1545968315583720. Epub 2015 Apr 20. PMID 25896988
- [Result] Chen S, Wolf SL, Zhang Q, Thompson PA, Winstein CJ. Minimal detectable change of the actual amount of use test and the motor activity log: the EXCITE Trial. Neurorehabil Neural Repair. 2012 Jun;26(5):507-14. doi: 10.1177/1545968311425048. Epub 2012 Jan 24. PMID 22275157
- [Result] Dusfour G, Mottet D, Muthalib M, Laffont I, Bakhti K. Comparison of wrist actimetry variables of paretic upper limb use in post stroke patients for ecological monitoring. J Neuroeng Rehabil. 2023 Apr 27;20(1):52. doi: 10.1186/s12984-023-01167-y. PMID 37106460
- [Result] Leuenberger K, Gonzenbach R, Wachter S, Luft A, Gassert R. A method to qualitatively assess arm use in stroke survivors in the home environment. Med Biol Eng Comput. 2017 Jan;55(1):141-150. doi: 10.1007/s11517-016-1496-7. Epub 2016 Apr 22. PMID 27106757
- [Result] Alt Murphy M, Willen C, Sunnerhagen KS. Kinematic variables quantifying upper-extremity performance after stroke during reaching and drinking from a glass. Neurorehabil Neural Repair. 2011 Jan;25(1):71-80. doi: 10.1177/1545968310370748. Epub 2010 Sep 9. PMID 20829411
- [Result] Noorkoiv M, Rodgers H, Price CI. Accelerometer measurement of upper extremity movement after stroke: a systematic review of clinical studies. J Neuroeng Rehabil. 2014 Oct 9;11:144. doi: 10.1186/1743-0003-11-144. PMID 25297823
- [Result] Platz T, Pinkowski C, van Wijck F, Kim IH, di Bella P, Johnson G. Reliability and validity of arm function assessment with standardized guidelines for the Fugl-Meyer Test, Action Research Arm Test and Box and Block Test: a multicentre study. Clin Rehabil. 2005 Jun;19(4):404-11. doi: 10.1191/0269215505cr832oa. PMID 15929509
- [Result] Saini V, Guada L, Yavagal DR. Global Epidemiology of Stroke and Access to Acute Ischemic Stroke Interventions. Neurology. 2021 Nov 16;97(20 Suppl 2):S6-S16. doi: 10.1212/WNL.0000000000012781. PMID 34785599
- [Result] Schambra HM, Parnandi A, Pandit NG, Uddin J, Wirtanen A, Nilsen DM. A Taxonomy of Functional Upper Extremity Motion. Front Neurol. 2019 Aug 20;10:857. doi: 10.3389/fneur.2019.00857. eCollection 2019. PMID 31481922
- [Result] Smith BA, Lang CE. Sensor Measures of Symmetry Quantify Upper Limb Movement in the Natural Environment Across the Lifespan. Arch Phys Med Rehabil. 2019 Jun;100(6):1176-1183. doi: 10.1016/j.apmr.2019.01.004. Epub 2019 Jan 29. PMID 30703350
- [Result] Sterr A, Freivogel S, Schmalohr D. Neurobehavioral aspects of recovery: assessment of the learned nonuse phenomenon in hemiparetic adolescents. Arch Phys Med Rehabil. 2002 Dec;83(12):1726-31. doi: 10.1053/apmr.2002.35660. PMID 12474177
- [Result] Stewart JC, Gordon J, Winstein CJ. Control of reach extent with the paretic and nonparetic arms after unilateral sensorimotor stroke: kinematic differences based on side of brain damage. Exp Brain Res. 2014 Jul;232(7):2407-19. doi: 10.1007/s00221-014-3938-5. Epub 2014 Apr 10. PMID 24718494
- [Result] Uswatte G, Hobbs Qadri L. A behavioral observation system for quantifying arm activity in daily life after stroke. Rehabil Psychol. 2009 Nov;54(4):398-403. doi: 10.1037/a0017501. PMID 19929121
- [Result] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Result] Zhou L, Fischer E, Tunca C, Brahms CM, Ersoy C, Granacher U, Arnrich B. How We Found Our IMU: Guidelines to IMU Selection and a Comparison of Seven IMUs for Pervasive Healthcare Applications. Sensors (Basel). 2020 Jul 22;20(15):4090. doi: 10.3390/s20154090. PMID 32707987
- [Result] Zou GY. Sample size formulas for estimating intraclass correlation coefficients with precision and assurance. Stat Med. 2012 Dec 20;31(29):3972-81. doi: 10.1002/sim.5466. Epub 2012 Jul 4. PMID 22764084